CLINICAL TRIAL: NCT00784576
Title: Incidence and Predictors of Delirium After Cardiac Surgery: A Prospective Observational Cohort Study
Brief Title: Incidence and Predictors of Delirium After Cardiac Surgery
Acronym: IPDACS
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Medical Universtity of Lodz, Poland, Medical Universtity of Lodz, Kosciuszki Street 4, 90-419 Lodz, Poland
Other Study IDs: 502-11-429
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-11

CONDITIONS: Delirium; Depression; Cognitive Impairment
Keywords: Delirium; Cardiac Surgery; Depression; Cognitive Impairment; Diagnostic Criteria for Delirium; Memorial Delirium Assessment Scale; Delirium Index
MeSH Terms: conditions — Delirium; Depression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery patients: Individuals consecutively scheduled for cardiac surgery

SUMMARY:
The objective of the present research is to evaluate the incidence and independent predictors of delirium observed among patients after cardiac surgery. Moreover, to asses the sensitivity and specificity of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criteria (DSM-IV) and International Statistical Classification of Diseases and Health Related Problems - Tenth Revision criteria (ICD-10), and the cut-off values of the Memorial Delirium Assessment Scale (MDAS) and Delirium Index (DI) in diagnosing postoperative delirium.

DETAILED DESCRIPTION:
Since 1954, the issue of delirium as a complication following cardiac surgery has been extensively investigated. Despite this, postoperative delirium is still a serious event that results in higher morbidity and mortality rates, and prolongs hospitalisation.

Moreover, there is a considerable discrepancy between studies on the incidence and risk factors of delirium among cardiac surgery patients.The first potential reason for this observation is retrospective design of some studies, secondly, the modest number of participants in numerous prospective studies which does not provide strong statistical power to select patients with delirium and detect risk factors of this complication. Unfortunately, reports with a more considerable number of patients often have methodological limitations. Additionally, in previous studies authors usually analyzed pre- and intraoperative variables ignoring potential postoperative risk factors of delirium. Finally, some variables which seem to have a crucial role in aetiology of delirium after cardiac surgery, particularly perioperative hypoxia, anaemia, and preoperative psychiatric disorders like depression and cognitive impairment, have not been properly investigated to date.

Therefore, we made an effort to design a prospective study on the incidence and predictors of delirium after different types of cardiac surgery, conducted by experienced investigators, and with the use of valid diagnostic tools.To our knowledge this is the first research pointing out the association between preoperative psychiatric comorbidity, anaemia and postoperative hypoxia, and delirium after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older
* Patients who signed an informed consent
* Patients scheduled for cardiac surgery with extracorporeal circulation (coronary-artery bypass grafting (CABG), cardiac valve replacement (CVR), combined CABG + CVR, excision of cardiac myxoma)

Exclusion Criteria:

* Patients who refuse to participate before or after operation
* Patients who undergo urgent surgery
* Patients in poor general condition
* Patients with preoperative dementia, delirium or illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of Cardiac Surgery in Lodz, Poland
Sampling Method: Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
MMSE and MINI - to assess cognitive performance and psychiatric comorbidity; DSM-IV and ICD-10 criteria; MDAS and DI - to estimate the incidence and severity of postoperative delirium; | one day before surgery; from the 2nd to the 6th day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Kazmierski, PhD, Principal Investigator — Department of Old-Age Psychiatry and Psychiatric Disorders, Medical University of Lodz, Poland; Maciej Banach, PhD, Study Director — Department of Cardiology, Medical University of Lodz, Poland
Locations (1):
- Department of Cardiac Surgery, 1st Chair of Cardiology and Cardiac Surgery, Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

REFERENCES:
- [Result] Kazmierski J, Kowman M, Banach M, Pawelczyk T, Okonski P, Iwaszkiewicz A, Zaslonka J, Sobow T, Kloszewska I. Preoperative predictors of delirium after cardiac surgery: a preliminary study. Gen Hosp Psychiatry. 2006 Nov-Dec;28(6):536-8. doi: 10.1016/j.genhosppsych.2006.08.007. PMID 17088170
- [Result] Kazmierski J, Sobow T, Kloszewska I. [Delirium after cardiac surgery]. Kardiol Pol. 2007 May;65(5):583-7. No abstract available. Polish. PMID 17577852
- [Result] Kazmierski J, Kowman M, Banach M, Fendler W, Okonski P, Banys A, Jaszewski R, Sobow T, Kloszewska I. Clinical utility and use of DSM-IV and ICD-10 Criteria and The Memorial Delirium Assessment Scale in establishing a diagnosis of delirium after cardiac surgery. Psychosomatics. 2008 Jan-Feb;49(1):73-6. doi: 10.1176/appi.psy.49.1.73. PMID 18212180
- [Result] Banach M, Kazmierski J, Kowman M, Okonski PK, Sobow T, Kloszewska I, Mikhailidis DP, Goch A, Banys A, Rysz J, Goch JH, Jaszewski R. Atrial fibrillation as a nonpsychiatric predictor of delirium after cardiac surgery: a pilot study. Med Sci Monit. 2008 May;14(5):CR286-291. PMID 18443554
- [Derived] Kazmierski J, Kowman M, Banach M, Fendler W, Okonski P, Banys A, Jaszewski R, Rysz J, Sobow T, Kloszewska I. The use of DSM-IV and ICD-10 criteria and diagnostic scales for delirium among cardiac surgery patients: results from the IPDACS study. J Neuropsychiatry Clin Neurosci. 2010 Fall;22(4):426-32. doi: 10.1176/jnp.2010.22.4.426. PMID 21037128
- [Derived] Kazmierski J, Kowman M, Banach M, Fendler W, Okonski P, Banys A, Jaszewski R, Rysz J, Mikhailidis DP, Sobow T, Kloszewska I; IPDACS Study. Incidence and predictors of delirium after cardiac surgery: Results from The IPDACS Study. J Psychosom Res. 2010 Aug;69(2):179-85. doi: 10.1016/j.jpsychores.2010.02.009. Epub 2010 Mar 30. PMID 20624517